CLINICAL TRIAL: NCT03525652
Title: Clinical Assessment of a Therapeutic Vaccine in Combination With PD-1 Knockout T Cells in the Treatment of Prostate Cancer
Brief Title: Therapeutic Vaccine Plus PD-1 Knockout in Prostate Cancer Treatment
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Guangdong Pharmaceutical University (Other)
Collaborators: Guangzhou Anjie Biomedical Technology Co., Ltd. (Industry); University of Technology, Sydney (Other)
Responsible Party: Principal Investigator, Size Chen, Professor, The First Affiliated Hospital of Guangdong Pharmaceutical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-007
Record Dates: First submitted 2018-04-26; First posted 2018-05-16 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Therapeutic vaccine; PD-1 knockout
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Therapeutic vaccine (Active Comparator): Therapeutic vaccine will be prepared ex vivo using the peripheral mononuclear cells from the patients and the vaccine (as maturated dendritic cells) will be infused back to the patients in 3 times with a 2-week interval.
  Interventions: Biological: Therapeutic vaccine
- Therapeutic vaccine plus PD-1 knockout (Experimental): Therapeutic vaccine and PD-1 knockout T cells will be prepared ex vivo using the white cells from the patients and the vaccine (as maturated dendritic cells) and maturated PD-1 knockout T cells will be infused back to the patients in 3 times.
  Interventions: Biological: Therapeutic vaccine; Biological: PD-1 Knockout T Cells
- PD-1 knockout T cells (Active Comparator): PD-1 knockout T cells will be prepared ex vivo using the white cells from the patients and the maturated PD-1 knockout T cells will be infused back to the patients in 3 times.
  Interventions: Biological: PD-1 Knockout T Cells

INTERVENTIONS:
Biological: Therapeutic vaccine — The therapeutic vaccine will be custom prepared ex vivo using the peripheral mononuclear cells from the patient and the vaccine which presented as maturated dendritic cells will be infused back to the patients in 3 times.
  Arms: Therapeutic vaccine; Therapeutic vaccine plus PD-1 knockout
Biological: PD-1 Knockout T Cells — PD-1 knockout T cells will be custom prepared ex vivo using the white blood cells from the patient and the maturated PD-1 knockout T cells will be infused back to the patients in 3 times.
  Arms: PD-1 knockout T cells; Therapeutic vaccine plus PD-1 knockout

SUMMARY:
This study is to evaluate the safety and efficacy of a therapeutic vaccine in combination with PD-1 knockout T cells in the treatment of advanced prostate cancer.

DETAILED DESCRIPTION:
This is a phase 1/2 clinical study investigating the safety and efficacy of a therapeutic vaccine in combination with PD-1 knockout T cells in the treatment of advanced prostate cancer. The therapeutic vaccine is a customized product involving ex vivo treatment of the patient's peripheral blood mononuclear cells with a recombinant fusion protein (PAP-GM-CSF) to activate the expression of the antigen that would activate the immune function to kill cancer cells. The PD-1 knockout engineered T cells are also prepared using patient's T cells in which PD-1 gene will be knocked out using CRISPR Cas9 technology. The therapeutic vaccine and PD-1 knockout T cells will be infused back to the patient in 3 times with a 2-week interval.

ELIGIBILITY:
Inclusion Criteria:

* • Histologically confirmed prostate cancer (stage IV, according to NCCN Clinical Practice Guidelines in Oncology: Prostate Cancer, Version 2.2017)

  * Evidence of metastasis in the soft tissue and/or bone.
  * Progressive androgen independent castrate resistant prostate cancer.
  * Serum PSA ≥ 5.0 ng/mL
  * Estimated life expectancy ≥ 6 months.
  * Castrate level of testosterone (< 50 ng/dL) achieved via medical or surgical castration.
  * Adequate hematologic, renal and liver function.

Exclusion Criteria:

* • Presence of known lung, liver, or brain metastases, malignant pleural effusions, or malignant ascites.

  * Presence of moderate to severe pain treating with opioid analgesics within 21 days prior to registration.
  * ECOG score ≥ 2.
  * Any other systemic therapy for prostate cancer (except for medical castration).
  * Participation in previous study using Provenge (Sipuleucel-T) or similar product.
  * Known pathologic long-bone fractures, imminent pathologic long-bone fracture (cortical erosion on radiography > 50%) or spinal cord compression.
  * Known malignancies other than prostate cancer requiring active treatment within 6 months.
  * A requirement for systemic immunosuppressive therapy for any reason.
  * A history of allergic reactions attributed to compounds of similar chemical or biologic composition to this product or granulocyte-macrophage colony-stimulating factor.
  * Any infection requiring parenteral antibiotic therapy or causing fever (temp > 100.5°F or > 38.1°C) within 1 week prior to registration.
  * Any medical intervention or other condition which, in the opinion of the Principal Investigator could compromise adherence with study requirements or otherwise compromise the study's objectives.
  * Treatment with any of the following medications or interventions within 28 days of registration:

Systemic use of corticosteroids, External beam radiation therapy or surgery, Use of non-steroidal antiandrogens Dietary and herbal supplements, as well as alternative treatments that have evidence of hormonal and/or anticancer properties (e.g., prostate cancer (PC) -SPES or PC-SPEC) and saw palmetto, Megestrol acetate (Megace®), diethylstilbesterol (DES), or cyproterone acetate, ++Ketoconazole, 5-alpha-reductase inhibitors, Treatment with any other investigational product Treatment with chemotherapy High dose calcitriol [1,25(OH)2Vitamin D] (i.e., > 0.5 mcg/day). Initiation or discontinuation of bisphosphonate therapy

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer is only presented in male
Enrollment: 30 (Estimated)
Dates: Start 2018-02-22 (Actual); Primary Completion 2021-02-22 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events and dose limiting toxicities as assessed by CTCAE v4.0 | 6 months
  Safety and tolerability of dose of therapeutic vaccine in combination with PD-1 Knockout T cells will be assessed using CTCAE v4.0

SECONDARY OUTCOMES:
Response Rate | 6 months
  Will be assessed according to the revised RECIST guideline v1.1
Progression free survival - PFS | Up to 12 months
  Time from treatment to date of first documented progression or date of death
Overall Survival - OS | Death
  Measure the time from the commencement of treatment to death
Peripheral blood circulating tumor DNA | 8 weeks
  Circuiting tumor DNA will be measured at baseline and 6 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Size Chen, MD, PhD, Principal Investigator — The First Affiliated Hospital of Guangdong Pharmaceutical University
Locations (2):
- China (2):
  - First Affiliated Hospital of Guangdong Pharmaceutical University, Guangzhou, Guangdong
  - Professor Size Chen, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No